CLINICAL TRIAL: NCT02874651
Title: ADjuVant Apatinib in Nasopharyngeal Carcinoma Patients With Residual Epstein-Barr Virus (EBV) DNA Following Radiotherapy With or Without Chemotherapy
Brief Title: ADjuVant Apatinib in Nasopharyngeal Carcinoma Patients With Residual Epstein-Barr Virus (EBV) DNA Following Radiotherapy
Acronym: ADVANCE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Unacceptable toxicity (nasopharynx necrosis and massive hemorrhage)
Sponsor: Sun Yat-sen University (Other)
Collaborators: First People's Hospital of Foshan (Other); Guilin Medical University, China (Other)
Responsible Party: Principal Investigator, Jun Ma, MD, Prof., Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Ahead-N301
Record Dates: First submitted 2016-08-01; First posted 2016-08-22 (Estimated); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Nasopharyngeal Neoplasms
Keywords: Nasopharyngeal Carcinoma; EB Virus; DNA; vascular endothecial growth factor receptor inhibitor; Apatinib
MeSH Terms: conditions — Nasopharyngeal Neoplasms; Nasopharyngeal Carcinoma; Epstein-Barr Virus Infections | interventions — apatinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Apatinib (Experimental): In the phase IIb part of this trial, patients in this arm will take oral apatinib until disease progression, intolerable toxicity, death or to a maximum of 2 years.
  Interventions: Drug: Apatinib
- Placebo (Placebo Comparator): In the phase IIb part of this trial, patients in this arm will take oral placebo until disease progression, intolerable toxicity, death or to a maximum of 2 years.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Apatinib — Patients will take oral apatinib. The initial dose is 500 mg once daily. 28 days as one cycle. After 1 cycle, the dose will be escalated to 750 mg once daily in patients with good tolerance. Dose interruption or reduction is permitted in case of adverse events per protocol.
  Other Names: YN968D1
  Arms: Apatinib
Drug: Placebo — Patients will take oral placebo. The initial dose is 500 mg once daily. 28 days as one cycle. After 1 cycle, the dose will be escalated to 750 mg once daily in patients with good tolerance. Dose interruption or reduction is permitted in case of adverse events per protocol.
  Other Names: Placebo tablet
  Arms: Placebo

SUMMARY:
This study will enroll patients with non-metastatic nasopharyngeal carcinoma (NPC) that have residual Epstein-Barr virus (EBV) DNA after curative radiotherapy or chemoradiotherapy. The purpose is to evaluate the survival in these patients treated with apatinib (YN968D1), an inhibitor of vascular endothelial growth factor receptor (phase IIa) and to compare the survival in these patients treated with apatinib versus placebo (phase IIb).

DETAILED DESCRIPTION:
This study has two parts. In the single arm phase IIa part, we will enroll 25 patients that have residual Epstein-Barr virus (EBV) DNA after curative radiotherapy or chemoradiotherapy. All patients will receive apatinib. The purpose is to evaluate the disease free-survival (DFS) in these patients treated with apatinib. In the phase IIb part, patients will be randomized to apatinib or placebo in a ratio of 1:1. The estimated sample size is 78 in phase IIb. However, the final sample size in phase IIb will be determined based on results of the phase IIa part.

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy proven nasopharyngeal carcinoma, with detectable pretreatment plasma EBV DNA
2. Have detectable plasma EBV DNA at the end of (+/- 1 week) curative radiotherapy or chemoradiotherapy (radiation dose > 66Gy), determined by the central lab
3. No clinical evidence of persistent loco-regional disease
4. No evidence of distant metastasis, based upon skeletal scintigraphy, chest X-ray examination, and liver ultrasound or other appropriate workup (e.g., CT, MRI or positron emission tomography (PET)/CT]) within 21 days prior to registration
5. Eastern Cooperative Oncology Group (ECOG) performance status 0-1
6. Anticipated survival >= 3 months
7. Absolute neutrophil count (ANC) >= 1,500 cells/mm^3
8. Platelets > 80,000 cells/mm^3
9. Hemoglobin >= 8.0 g/dl (no transfusion within the last 14 days)
10. Total bilirubin =< 1.5 x institutional upper limit of normal (ULN)
11. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) =< 2.5 x institutional ULN
12. Creatinine clearance (CC) >= 50 ml/min estimated by Cockcroft-Gault formula

Exclusion Criteria:

1. Patients with stage III-IV disease (American Joint Committee On Cancer/Union for International Cancer Control 7th) and no contraindication to chemotherapy that didn't receive platinum based concurrent chemotherapy during radiation
2. Patients with tumor possibly invaded main vessels (e.g. encasement of the internal jugular artery/vein) at diagnosis; or tumor that, in the judgment of the investigator, likely to invade main vessels and cause life-threatening hemorrhage events during study
3. History of serious hemorrhage events or grade 3 or higher hemorrhage within 4 weeks prior to registration
4. Hypertension that couldn't be well controlled with single medication; unstable angina; angina diagnosed within the last 3 months; myocardial infarction within the last 6 months; cardiac arrhythmia that need long-term medication; grade 2 or higher cardiac dysfunction (NYHA)
5. Proteinuria
6. Coagulation dysfunction or predisposition to hemorrhage; on treatment of anticoagulation medication or vitamin K antagonist; low dose warfarin (1mg po qd) or aspirin (less than 100mg daily) were permitted as long as the international normalized ratio (INR) = < 1.5
7. Thrombosis within the last 1 year, except cured vein thrombosis related to vein indwelling catheter
8. Unhealed bone fracture or chronic unhealed wound
9. Illness that would interfere with oral medication, including dysphagia, chronic diarrhea, or ileus
10. Pregnant or lactating women
11. Women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception during and within 6 months after study
12. Current drug abuse or mentally disabled
13. History of congenital or acquired immune deficiency disease or organ transplantation
14. Major medical illness, which in the investigator's opinion would endanger the patients or interfere with the completion of therapy and follow up

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-10; Primary Completion 2018-11-29 (Actual); Study Completion 2020-08-27 (Actual)

PRIMARY OUTCOMES:
Disease-free survival | 3 years

SECONDARY OUTCOMES:
overall survival | 5 years
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 2 years
Changes in quality of life (QOL) as assessed by EORTC QLQ-C30 | 2 years
Distance Metastasis Free Survival | 3 years
locoregional relapse free survival | 3 years
Correlation of plasma EBV DNA load with the effect of apatinib on survival | 3 years
Correlation of pretreatment serum VEGF level with the effect of apatinib on survival | 3 years
Correlation of pretreatment serum VEGFR-2 level with the effect of apatinib on survival | 3 years
Correlation of adverse event (hypertension) with the effect of apatinib on survival | 3 years
Correlation of adverse event (hand-foot syndrome) with the effect of apatinib on survival | 3 years
Correlation of the change from baseline in serum VEGF level at 4 weeks with the effect of apatinib on survival | 3 years
Correlation of the change from baseline in serum VEGFR-2 level at 4 weeks with the effect of apatinib on survival | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jun Ma, M.D., Study Chair — Sun Yat-sen University
Locations (3):
- China (3):
  - Affiliated Foshan Hospital of Sun Yat-sen University, Foshan, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Affiliated Hospital of Guilin Medical University, Guilin, Guangxi

IPD SHARING:
Plan to Share IPD: No